CLINICAL TRIAL: NCT01591317
Title: Single and Multiple Dose Pharmacokinetics and Pharmacodynamics of Prasugrel (LY640315) in Korean Healthy Male Subjects
Brief Title: Study of Prasugrel in Korean Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11990; H7T-FW-TACQ (Other: Eli Lilly and Company)
Record Dates: First submitted 2012-05-02; First posted 2012-05-04 (Estimated); Results first posted 2012-10-04 (Estimated); Last update posted 2012-10-04 (Estimated); Status verified 2012-09

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Prasugrel Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Prasugrel - 60 mg/10 mg (Experimental): Prasugrel 60 mg loading dose given once orally, followed by 10 mg once a day orally for 10 days
  Interventions: Drug: Prasugrel
- Prasugrel - 30 mg/7.5 mg (Experimental): Prasugrel 30 mg loading dose given once orally, followed by 7.5 mg once a day orally for 10 days
  Interventions: Drug: Prasugrel
- Prasugrel - 30 mg/5 mg (Experimental): Prasugrel 30 mg loading dose given once orally followed by 5 mg once a day orally for 10 days
  Interventions: Drug: Prasugrel

INTERVENTIONS:
Drug: Prasugrel — Tablets orally
  Other Names: LY640315; Effient; Efient; Prasita

SUMMARY:
The purpose of this study is to investigate how the body processes prasugrel and how prasugrel affects blood clotting in healthy Korean men. Three different dosing regimens of prasugrel will be given. Information on side effects will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy males, as determined by medical history and physical examination.
* Are between the ages of 20 and 45 years, inclusive.
* Have a body mass index (BMI) of 19 kg/m^2 to 27 kg/m^2, inclusive, at screening.

Exclusion Criteria:

* Are currently enrolled in, or discontinued within the last 60 days from a clinical trial involving an investigational drug or device, or are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study.
* Have known allergies to prasugrel or related compounds.
* Are persons who have previously completed or withdrawn from this study or any other study investigating prasugrel.
* Self-reported history of significant bleeding from trauma (for example, prolonged bleeding after tooth extraction).
* History of major surgery within 3 months of screening or planned surgery within 14 days after the last day of dosing.
* Have a platelet count of <100,000/(cubic millimeters) mm^3 at the time of screening.
* Have tested positive for fecal occult blood at screening.
* Have significant prolongation of prothrombin time (PT) or activated partial thromboplastin time (APTT) at screening.
* Have a clinically significant abnormality following the investigator's review of the physical examination, electrocardiogram (ECG)and clinical (safety) laboratory tests at screening.
* Personal or first-degree family history of coagulation or bleeding disorders (that is, hematemesis, melena, severe or recurrent epistaxis, hemoptysis, gastrointestinal ulcers, hemorrhage, clinically overt hematuria or intracranial hemorrhage) or reasonable suspicion of vascular malformations, for example, cerebral hemorrhage, aneurysm or premature stroke (cerebrovascular accident [CVA] <65 years of age).
* Have significant active hematological disease and/or whole blood donation of more than 400 mL within the last 2 months and component blood donation within the last month.
* Volunteers who have an average weekly alcohol intake that exceeds 21 units per week or volunteers unwilling to adhere to study alcohol restrictions during the study (1 unit = 360 mL of beer; 150 mL of wine; 45 mL of distilled spirits).

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2009-03; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seoul, South Korea

REFERENCES:
- [Derived] Yu KS, Park KW, Kelly RP, Gu N, Payne C, Small DS, Choi HC, Kawakatsu E, Pinton P. Pharmacokinetic and pharmacodynamic effects of prasugrel in healthy Korean males. J Cardiovasc Pharmacol. 2013 Jul;62(1):72-7. doi: 10.1097/FJC.0b013e318290d9e1. PMID 23594968

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Prasugrel - 60 mg/10 mg | Prasugrel - 30 mg/7.5 mg | Prasugrel - 30 mg/5 mg
Started | 10 | 10 | 10
Completed | 10 | 10 | 10
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prasugrel - 60 mg/10 mg | Prasugrel - 30 mg/7.5 mg | Prasugrel - 30 mg/5 mg | Total
Number analyzed (Participants) | 10 | 10 | 10 | 30
Age Continuous [Mean (Standard Deviation); unit: years] | 28.2 (5.3) | 25.9 (5.2) | 26.0 (4.1) | 26.7 (4.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 10 | 10 | 10 | 30
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 10 | 10 | 10 | 30
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 10 | 10 | 10 | 30

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Area Under the Concentration Curve (AUC) of Prasugrel's Active Metabolite R-138727 During Loading Dose
Description: AUC from time zero to the last quantifiable plasma concentration (tlast)
Time Frame: Day 1 predose up to 24 hours post dose
Population: All randomized participants
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram times hour/milliliter (ng*h/mL)
Groups:
- Prasugrel 60 mg: Prasugrel 60 mg loading dose given once orally
- Prasugrel 30 mg: Prasugrel 30 mg loading dose given once orally
Arm/Group | Prasugrel 60 mg | Prasugrel 30 mg
Number analyzed (Participants) | 10 | 20
nanogram times hour/milliliter (ng*h/mL) | 600 (16) | 283 (17)

2. Primary Outcome: Pharmacokinetics (PK): Maximum Concentration (Cmax) for Prasugrel's Active Metabolite R-138727 During Loading Dose
Time Frame: Day 1 predose up to 24 hours post dose
Population: All randomized participants
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/milliliter (ng/mL)
Arm/Group | Prasugrel 60 mg | Prasugrel 30 mg
Number analyzed (Participants) | 10 | 20
nanogram/milliliter (ng/mL) | 498 (41) | 271 (39)

3. Primary Outcome: Pharmacokinetics (PK): Time to Maximum Concentration (Tmax) of Prasugrel's Active Metabolite R-138727 During Loading Dose
Time Frame: Day 1 predose up to 24 hours post dose
Population: All randomized participants
Measure: Median (Full Range); unit: hours
Arm/Group | Prasugrel 60 mg | Prasugrel 30 mg
Number analyzed (Participants) | 10 | 20
hours | 0.50 [0.25 to 1.00] | 0.50 [0.25 to 1.00]

4. Secondary Outcome: Pharmacodynamics: Adenosine Diphosphate (ADP)-Induced P2Y12 Receptor-mediated Platelet Aggregation
Description: ADP-induced PRU represents the rate and extent of ADP-stimulated platelet aggregation and serves as a biomarker of clinical efficacy, with lower values indicating greater P2Y12 platelet inhibition
Time Frame: Predose up to 24 hours post dose on Day 12
Population: All randomized participants
Measure: Mean (Standard Deviation); unit: PRU
Arm/Group | Prasugrel - 60 mg/10 mg | Prasugrel - 30 mg/7.5 mg | Prasugrel - 30 mg/5 mg
Number analyzed (Participants) | 10 | 10 | 10
PRU
  Day 1, predose | 290 (36.2) | 273 (39.6) | 297 (48.9)
  Day 1, 0.5 hours | 118 (120) | 107 (95.5) | 172 (102)
  Day 1, 1 hour | 13.5 (18.9) | 19.0 (42.6) | 46.0 (45.0)
  Day1, 2 hours | 3.30 (2.16) | 7.00 (11.3) | 20.1 (29.0)
  Day 1, 4 hours | 2.70 (1.89) | 3.10 (1.73) | 12.1 (24.0)
  Day 1, 24 hours | 7.10 (9.52) | 5.10 (2.56) | 26.9 (32.2)
  Day 10, predose | 34.8 (51.4) | 35.1 (25.0) | 121 (53.7)
  Day 11, predose | 39.6 (61.9) | 26.4 (27.7) | 123 (45.8)
  Day 11, 24 hours | 24.4 (26.7) | 27.2 (31.8) | 107 (53.7)

5. Primary Outcome: Pharmacokinetics (PK): Area Under the Concentration Curve (AUC) of Prasugrel's Active Metabolite R-138727 During Maintenance Dose
Description: AUC from time zero to the last quantifiable plasma concentration (tlast)
Time Frame: Day 11 predose to 24 hours post dose
Population: All randomized participants
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- Prasugrel 10 mg: Prasugrel 10 mg once a day orally for 10 days
- Prasugrel 7.5 mg: Prasugrel 7.5 mg once a day orally for 10 days
- Prasugrel 5 mg: Prasugrel 5 mg once a day orally for 10 days
Arm/Group | Prasugrel 10 mg | Prasugrel 7.5 mg | Prasugrel 5 mg
Number analyzed (Participants) | 10 | 10 | 10
ng*h/mL | 78.1 (24) | 58.4 (21) | 38.3 (24)

6. Primary Outcome: Pharmacokinetics (PK): Maximum Concentration (Cmax) for Prasugrel's Active Metabolite R-138727 During Maintenance Dose
Time Frame: Day 11 predose to 24 hours post dose
Population: All randomized participants
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Prasugrel 10 mg | Prasugrel 7.5 mg | Prasugrel 5 mg
Number analyzed (Participants) | 10 | 10 | 10
ng/mL | 92.3 (36) | 61.9 (37) | 41.0 (73)

7. Primary Outcome: Pharmacokinetics (PK): Time to Maximum Concentration (Tmax) of Prasugrel's Active Metabolite R-138727 During Maintenance Dose
Time Frame: Day 11 predose to 24 hours post dose
Population: All randomized participants
Measure: Median (Full Range); unit: hours
Arm/Group | Prasugrel 10 mg | Prasugrel 7.5 mg | Prasugrel 5 mg
Number analyzed (Participants) | 10 | 10 | 10
hours | 0.50 [0.25 to 0.50] | 0.50 [0.25 to 0.52] | 0.38 [0.25 to 1.00]

8. Secondary Outcome: Percent Inhibition of Verify Now (VN)-P2Y12 Reaction Units (PRU)
Description: PRU device reported VerifyNow percent inhibition is reported by Accumetrics VerifyNow™ P2Y12 (VN-P2Y12) assay, a point-of-care device that measures platelet aggregation with single-use, disposable cartridges
Time Frame: Predose up to 24 hours post dose on Day 12
Population: All randomized participants
Measure: Mean (Standard Deviation); unit: Percent inhibition of PRU
Arm/Group | Prasugrel - 60 mg/10 mg | Prasugrel - 30 mg/7.5 mg | Prasugrel - 30 mg/5 mg
Number analyzed (Participants) | 10 | 10 | 10
Percent inhibition of PRU
  Day 1, predose | 9.90 (10.9) | 6.80 (5.57) | 9.90 (11.4)
  Day 1, 0.5 hours | 64.9 (35.5) | 66.9 (28.9) | 48.8 (29.2)
  Day 1, 1 hour | 95.8 (6.00) | 94.2 (13.9) | 86.9 (12.3)
  Day1, 2 hours | 98.9 (0.568) | 97.7 (3.47) | 94.0 (8.26)
  Day 1, 4 hours | 99.2 (0.632) | 99.1 (0.738) | 96.8 (6.00)
  Day 1, 24 hours | 97.8 (2.94) | 98.3 (0.675) | 92.0 (9.51)
  Day 10, predose | 89.3 (15.7) | 87.6 (8.82) | 63.6 (14.7)
  Day 11, predose | 88.5 (18.4) | 91.2 (9.07) | 64.8 (12.9)
  Day 11, 24 hours | 92.5 (7.43) | 91.0 (10.0) | 67.0 (17.2)

ADVERSE EVENTS:
Arm/Group | Prasugrel - 60 mg/10 mg | Prasugrel - 30 mg/7.5 mg | Prasugrel - 30 mg/5 mg
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 3/10 | 4/10 | 3/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prasugrel - 60 mg/10 mg (N=10) | Prasugrel - 30 mg/7.5 mg (N=10) | Prasugrel - 30 mg/5 mg (N=10)
Chest discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0)
Vessel puncture site paraesthesia (General disorders) | 1 (1) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Sputum retention (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days